CLINICAL TRIAL: NCT06999590
Title: A Multicenter, Prospective, Randomized Controlled Modified Platform Trial Evaluating Several Cellular, Acellular, and Matrixlike Products (CAMPs) and Standard of Care Versus Matched Standard of Care Controls in the Management of Nonhealing Pressure Ulcers
Brief Title: Evaluating Several Cellular, Acellular, and Matrix-like Products (CAMPs) and Standard of Care Versus Matched Standard of Care Controls in the Management of Nonhealing Pressure Ulcers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tiger Biosciences, LLC. (Industry)
Collaborators: ExtremityCare, LLC. (Unknown); SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIGERTAIL
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pressure Ulcer; Ulcer; Ulcer, Pressure; Pressure Injury
MeSH Terms: conditions — Pressure Ulcer; Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective Modified Platform Multicenter Clinical Trial Utilizing Matched Controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACApatch™ + SOC (Experimental): Human amniotic membrane tissue allografts derived from human placental tissue.
  Interventions: Other: ACApatch™
- caregraFT™ + SOC (Experimental): Human amniotic membrane tissue allografts derived from human placental tissue.
  Interventions: Other: caregraFT™
- Standard of Care (Active Comparator): Standard of care will be cleaning, debridement, and ulcer moisture balance.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: ACApatch™ — Participants will receive weekly applications of ACApatch™ and Standard of Care until ulcer closure, or a maximum of 20 weeks, whichever occurs first.
  Arms: ACApatch™ + SOC
Other: caregraFT™ — Participants will receive weekly applications of caregraFT™ and Standard of Care until ulcer closure, or a maximum of 20 weeks, whichever occurs first.
  Arms: caregraFT™ + SOC
Other: Standard of Care — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance) until ulcer closure, or a maximum of 20 weeks, whichever occurs first.
  Arms: Standard of Care

SUMMARY:
The purpose of this study it to evaluate several cellular, acellular, and matrix-like products (CAMPs) and standard of care versus matched standard of care controls in the management of nonhealing pressure ulcers.

DETAILED DESCRIPTION:
To determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing pressure ulcers with multiple CAMPs plus SOC versus matched SOC controls (mSOC) over 20 weeks using a modified platform trial design. The initial plan is to evaluate two CAMPs; however, the modified platform design permits the inclusion of additional CAMPs.

ELIGIBILITY:
Inclusion Criteria:

1. The potential subject must be at least 18 years of age or older.
2. The potential subject must agree to attend the weekly study visits required by the protocol.
3. The potential subject must be willing and able to participate in the informed consent process.
4. The potential subject must have a full-thickness pressure ulcer NPIAP stage 3 or stage 4 without exposed tendon or bone of greater than or equal to one month in duration located on the trunk (sacral, trochanteric, or ischial).
5. At enrollment, the potential subject must have a target ulcer with a minimum surface area of 2 cm2 and a maximum surface area of 100 cm2 measured post-debridement with the imaging device.
6. The potential subject has adequate off-loading of the ulcer.

Exclusion Criteria:

1. The potential subject is known to have a life expectancy of < 3 months.
2. The potential subject's target ulcer is not a pressure ulcer.
3. The target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
4. The target ulcer exposes tendon or bone.
5. The target ulcer has undermining or tunneling.
6. There is evidence of osteomyelitis complicating the target ulcer.
7. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
8. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
9. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
10. The surface area of the potential subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
11. The surface area measurement of the potential subject's target ulcer decreases by 25% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1 visit during which time the potential subject received SOC.
12. The potential subject is a woman who is pregnant or considering becoming pregnant within the next 6 months.
13. The potential subject has end stage renal disease requiring dialysis.
14. The potential subject, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
15. The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
16. The potential subject has a malnutrition indicator score of <17 as measured on the Mini Nutritional Assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Complete closure | 1-20 Weeks
  To determine the between-arm difference in the proportion of subjects achieving complete closure of nonhealing pressure ulcers with multiple CAMPs plus SOC versus matched SOC controls (mSOC) over 20 weeks using a modified platform trial design.

SECONDARY OUTCOMES:
Time to Closure | 1-20 weeks
  To determine the between-arm difference in the time to closure over 16 weeks for CAMP plus SOC versus mSOC.
Percentage Area Reduction | 1-20 weeks
  To determine the between-arm difference in the percent area reduction (PAR) at weekly intervals the CAMP plus SOC arms versus mSOC.
Determine Quality of Life | 1-20 weeks
  To determine the between-arm difference in pain for patients that present with a VAS score of greater than 4. Pain will be rated on a scale of 0 to 10, with 0 meaning no pain and 10 meaning the most pain.
Adverse Events | 1-20 weeks
  To evaluate the between-arm difference in the frequency and nature of adverse events in subjects receiving CAMP plus SOC versus mSOC.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD, Principal Investigator — Serena Group
Locations (1):
- Serena Group, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No